CLINICAL TRIAL: NCT04946058
Title: Hybrid Mathieu Urethroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mohammad Gharieb Mohammad Khirallah, Assistant professor of pediatric surgery, Tanta University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 34403//1/21
Record Dates: First submitted 2021-06-16; First posted 2021-06-30 (Actual); Last update posted 2021-06-30 (Actual); Status verified 2021-06

CONDITIONS: Distal Penile Hypospadias (Disorder)
Keywords: distal hypospadias; Mathieu urethroplasty; modified; urethral plate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: hyebrid Mathieu Urethroplasty — incision of the urethral plate during the procedure

SUMMARY:
the aim is to study the results of simple modification of classic Mathieu urethroplasty to increase the scope of cases candidates for that procedure.

DETAILED DESCRIPTION:
background: Distal hypospadias repair is one of most frequent surgical interventions in pediatric age group. Successful hypospadias repair should provide a functional penis and good cosmesis. Mathieu urethroplasty is one of the most popular techniques used. Authors aimed at performing a modification that expanded the scope of indications and improved final cosmetic results of classic Mathieu urethroplasty.

Methods: forty-three patients with distal hypospadias were operated by hybrid Mathieu urethroplasty (HMU) during the period from March 2012 to December 2020. Creation of the peri meatal based flap was performed as Mathieu disrobed. This was followed by developing of glanular wings. The additional step was deep incision of the urethral plate. Then, urethroplasty was performed. The catheter was left in place for one to three days.

ELIGIBILITY:
Inclusion Criteria:

* distal penile hypospadias

Exclusion Criteria:

* sever hypospadias
* cases need redo

Ages: 6 Months to 4 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes — all male infants and children suffering from distal penile hypospadias
Enrollment: 43 (Actual)
Dates: Start 2012-03-31 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-01-15 (Actual)

PRIMARY OUTCOMES:
successful treatment of distal penile hypospadias | 6 moths post operative
  use of HOSE as a measure o success o repair
increase the scope of classic Mathieu urethroplasty | 6 months post operative
  cases with glanular width from 10 mm to 15 mm were included

IPD SHARING:
Plan to Share IPD: Undecided
publishing an article including the operative details and results